CLINICAL TRIAL: NCT03405506
Title: Functional Diagnostic Accuracy of Quantitative Flow Ratio in Tandem Lesions and Virtual Stenting
Acronym: FORTRESS
Status: Completed | Type: Observational
Sponsor: Pulse Medical Imaging Technology (Shanghai) Co., Ltd (Industry)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIAC201701
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases; Myocardial Ischemia; Arterial Occlusive Diseases; Heart Diseases; Vascular Diseases; Arteriosclerosis
Keywords: Fractional Flow Reserve; Quantitative Coronary Angiography; Coronary artery disease; Quantitative Flow Ratio; Tandem lesion; Virtual stenting
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Myocardial Ischemia; Arterial Occlusive Diseases; Heart Diseases; Vascular Diseases; Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Quantitative Flow Ratio (QFR) — FFR measured by pressure wire, QFR computed by coronary angiographic images

SUMMARY:
Quantitative Flow Ratio (QFR) is a novel method for evaluating the functional significance of coronary stenosis. Virtual stent implantation technique combined with QFR was recently developed to predict the functional significance of coronary stenosis as if the stenosis was revascularized.

The purpose of this study is to evaluate the diagnostic accuracy of QFR in in tandem lesions with fractional flow reserve (FFR) as the reference standard. The secondary purpose is to evaluate the diagnostic accuracy of QFR-based virtual stent technique in predicting the FFR values after revascularizing the culprit lesion.

DETAILED DESCRIPTION:
QFR is a novel method for evaluating the functional significance of coronary stenosis by calculation of the pressure drop in the vessel. 3D coronary models can be reconstructed based on two angiographic projections to obtain the geometric parameters, including vascular diameter or cross-sectional area. According to the lesion stenosis, vessel curvature, conical geometry and reference lumen characteristics, pressure drop can be calculated in real time based on its relationship with blood flow. There is no need for pressure wire and adenosine / ATP induced maximum hyperemia compared with FFR.

The FAVOR Pilot Study and FAVOR II China Study showed promising results for diagnostic accuracy in consecutive patients. However, the diagnostic accuracy of QFR in specific tandem lesions needs further investigation. Furthermore, using the virtual stent technology to accurately assess the culprit lesion and choose the optimal treatment is significant in precisely guiding PCI surgery.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion Criteria:

  1. Stable and unstable angina pectoris or secondary evaluation of stenosis after acute MI;
  2. Age > 18 years;
  3. Able to provide signed informed consent.
* Angiographic inclusion criteria:

  1. At least two localized lesions on the same coronary artery;
  2. More than 50% diameter stenosis (DS) estimated by QCA on each lesion;
  3. At least 10 mm relatively normal lumen (at most 20% DS) between two lesions;
  4. Reference vessel size > 2 mm in stenotic segment by visual estimate.

Exclusion Criteria:

* General exclusion criteria:

  1. Ineligible for diagnostic intervention or FFR examination;
  2. Myocardial infarction within 72 hours;
  3. Severe heart failure (NYHA≥III);
  4. S-creatinine>150µmol/L or GFR<45 ml/kg/1.73m2;
  5. Allergy to contrast agent or adenosine;
  6. Factors that might substantially impact the angiographic image quality, e.g, frequent atrial premature beat or atrial fibrillation;
  7. Serious complications:

     1. Evidence of cardiac rupture;
     2. History of bleeding (intracranial hemorrhage, gastrointestinal bleeding, etc.);
     3. Acute or chronic blood system diseases, including hemoglobin < 10 g / L, or platelet count < 50 × 109 / L;
     4. Accompanied by other diseases might inducing life expectancy shorter than several months;
     5. History of severe renal insufficiency and hypohepatia (liver failure, cirrhosis, portal hypertension and active hepatitis)
     6. Aneurysm, arterial / venous malformation, aortic dissection;
  8. Cardiogenic shock or circulation capacity failure;
  9. Two-degree and more severe atrioventricular block, with no permanent pacemaker implanted;
  10. Pregnancy or lactation;
  11. The investigators believe that the treatment regimen may be detrimental to the patient or the enrollment of this subject may affect the specific assessment of the trial;
* Angiographic exclusion criteria:

  1. The interrogated stenosis is caused by myocardial bridge;
  2. Ostial lesions less than 3 mm to the aorta;
  3. Side branches of the bifurcation lesions with Median Classification of 111 or 101;
  4. Severe overlap or shorten of stenosis segment;
  5. Severe tortuosity of target vessel;
  6. Poor angiographic image quality precluding contour detection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary tandem lesions admitted for coronary angiography due to high risk of significant coronary stenosis
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of QFR in tandem lesions as compared with FFR prior to intervention | 1 hour
  Diagnostic accuracy was defined as the concordance ratio of QFR evaluated outcomes (≤ 0.8 or > 0.8) with the reference standard FFR evaluated outcomes (≤ 0.8 or > 0.8)

SECONDARY OUTCOMES:
Diagnostic accuracy of QFR-based virtual stenting in predicting FFR values after revascularizing the culprit lesion | 1 hour
  Diagnostic accuracy was defined as the concordance ratio of QFR evaluated outcomes (≤ 0.8 or > 0.8) with the reference standard FFR evaluated outcomes (≤ 0.8 or > 0.8)

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739